CLINICAL TRIAL: NCT06802185
Title: A Randomized, Open Label, Single Oral Dose, Four Treatment, Four Period, Four Sequence, Crossover Bioequivalence Study of Advil Dual Action Liquid Filled Capsules (125 mg/250 mg) vs Advil Dual Action Caplets (125 mg/250 mg) in Healthy Adult Subjects Under Fasted Conditions, and Bioavailability Assessment of Advil Dual Action Liquid Filled Capsules (125 mg/250 mg) Under Fed Conditions and Advil Liqui-Gels (200 mg) Under Fasted Conditions
Brief Title: A Bioequivalence Study of Advil Dual Action Liquid Filled Capsules (125 mg/250 mg) Versus Advil Dual Action Caplets (125 mg/250 mg) and Bioavailability Assessment of Advil Dual Action Liquid Filled Capsules (125 mg/250 mg) and Advil Liqui-Gels (200 mg) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 300219
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1: Treatment A + Treatment B + Treatment C + Treatment D (Experimental): Participants will receive a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 1 (Treatment A), followed by a single oral dose of 2 ADA Caplets (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 2 (Treatment B), followed by a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fed conditions, 30 minutes after a high-fat high calorie meal on Day 1 of Period 3 (Treatment C) and further followed by a single oral dose of 2 Advil Liqui-gels (ibuprofen 200 mg) under fasted conditions on Day 1 of Period 4 (Treatment D). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: ADA Liquid Filled Capsules (Test Product); Drug: ADA Caplets (Reference Product); Drug: Advil Liqui-gels (Reference Product)
- Sequence 2: Treatment B + Treatment D + Treatment A + Treatment C (Experimental): Participants will receive a single oral dose of 2 ADA Caplets (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 1 (Treatment B), followed by a single oral dose of 2 Advil Liqui-gels (ibuprofen 200 mg) under fasted conditions on Day 1 of Period 2 (Treatment D), followed by a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 3 (Treatment A) and further followed by a single oral dose of ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fed conditions, 30 minutes after a high-fat high calorie meal on Day 1 of Period 4 (Treatment C). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: ADA Liquid Filled Capsules (Test Product); Drug: ADA Caplets (Reference Product); Drug: Advil Liqui-gels (Reference Product)
- Sequence 3: Treatment C + Treatment A + Treatment D + Treatment B (Experimental): Participants will receive a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fed conditions, 30 minutes after a high-fat high calorie meal on Day 1 of Period 1 (Treatment C), followed by a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 2 (Treatment A), followed by a single oral dose of 2 Advil Liqui-gels (ibuprofen 200 mg) under fasted conditions on Day 1 of Period 3 (Treatment D) and further followed by a single oral dose of 2 ADA Caplets (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 4 (Treatment B). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: ADA Liquid Filled Capsules (Test Product); Drug: ADA Caplets (Reference Product); Drug: Advil Liqui-gels (Reference Product)
- Sequence 4: Treatment D + Treatment C + Treatment B + Treatment A (Experimental): Participants will receive a single oral dose of 2 Advil Liqui-gels (ibuprofen 200 mg) under fasted conditions on Day 1 of Period 1 (Treatment D), followed by a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fed conditions, 30 minutes after a high-fat high calorie meal on Day 1 of Period 2 (Treatment C), followed by a single oral dose of 2 ADA Caplets (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 3 (Treatment B), and further followed by a single oral dose of 2 ADA liquid filled capsules (125 mg ibuprofen and 250 mg acetaminophen) under fasted conditions on Day 1 of Period 4 (Treatment A). There will be a washout period of at least 3 days between each treatment.
  Interventions: Drug: ADA Liquid Filled Capsules (Test Product); Drug: ADA Caplets (Reference Product); Drug: Advil Liqui-gels (Reference Product)

INTERVENTIONS:
Drug: ADA Liquid Filled Capsules (Test Product) — ADA liquid filled capsules containing 125 mg ibuprofen and 250 mg acetaminophen.
Drug: ADA Caplets (Reference Product) — ADA Caplets containing 125 mg ibuprofen and 250 mg acetaminophen.
Drug: Advil Liqui-gels (Reference Product) — Advil Liqui-gels containing 200 mg ibuprofen.

SUMMARY:
The primary purpose of this study is to demonstrate the bioequivalence of new formulation Advil Dual Action (ADA) liquid filled capsules (Test) compared to the currently marketed ADA Caplet (Reference) under fasted conditions and to assess the relative bioavailability of ADA liquid filled capsules (Test) under fed conditions compared to ADA liquid filled capsules (Reference) under fasted conditions.

DETAILED DESCRIPTION:
This is a single center, single oral dose, open-label, randomized, four-treatment, four period, four sequence, crossover, bioequivalence study of ADA liquid filled capsules (125 milligrams [mg] ibuprofen/250 mg acetaminophen) (Treatment A) versus (vs.) ADA Caplets (125 mg ibuprofen/250 mg acetaminophen) (Treatment B) in healthy adult participants under fasted conditions. The study also includes a bioavailability assessment of ADA liquid filled capsules (125 mg ibuprofen/250 mg acetaminophen) under fed conditions (Treatment C) and Advil Liqui-Gels (200 mg ibuprofen) under fasted conditions (Treatment D). A sufficient number of male and female participants will be screened to randomize approximately 54 to ensure at least 48 evaluable participants complete the entire study. Participants will be randomly assigned to 1 of the 4 treatment sequences and receive a single oral dose of the investigational products per the randomization in each period following a crossover design. There will be a wash-out period of 3 days between investigational product administrations. Blood will be sampled regularly at scheduled times for 24 hours following treatment in each period to assess the pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is male or female who, at the time of screening, is between the ages of 18 and 55 years, inclusive. An effort will be made to include similar proportions of males and females in the study.
* Participant who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon the physical examination, blood pressure (BP) and pulse rate measurement, 12-lead electrocardiogram (ECG) or clinical laboratory tests, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the participant's ability to understand and follow study procedures and requirements.
* Body Mass Index (BMI) of 18.5 to 30.0 kilogram per meter square (kg/m^2); and a total body weight more than or equal to (>=) 50.0 kilograms (kg) for males and >= 45.0 kg for females at screening.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or intends to participate in any other study during participation in this study.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Pregnant female participant as confirmed by a positive pregnancy test or intending to become pregnant over the duration of the study.
* Breastfeeding female participant.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Any history of asthma, urticaria, or other significant allergic diathesis or allergic reaction to any other pain reliever/fever reducer. Participant with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly outside enrollment/treatment period.
* Diagnosis of long QT syndrome or QT corrected for heart rate by Fridericia's cube root formula (QTcF) more than (>) 450 milliseconds (msec) for males and >470 msec for females at screening.
* Vital sign abnormalities (systolic BP lower than 90 or over 140 millimeters of mercury (mmHg), diastolic BP lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 beats per minute) unless determined by the Investigator or medically qualified designee to be not clinically significant. Vital signs may be repeated at the discretion of the Investigator or medically qualified designee.
* Unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* Use of any medication (including over the counter medications and herbal remedies) within 2 weeks or within less than 10 times the elimination half-life of the respective drug (whichever is longer) before first scheduled study drug administration, or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  1. systemic contraceptives as long as female participant is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study.
* Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease in the opinion of the Investigator, or medically qualified designee that may increase the risk associated with study participation.
* Any history of long-term treatment with carbamazepine, phenobarbitone, phenytoin, primidone, rifampicin, St John's Wort or other drugs that induce liver enzymes.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to start of the study.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance including, but not limited to any of the following:

  1. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, example, appendectomy and herniorrhaphy);
  2. History of inflammatory bowel disease or gastrointestinal bleeding including peptic ulcers;
  3. History or current evidence of renal disease or impaired renal function at screening as demonstrated by an estimated glomerular filtration rate (eGFR) less than (<) 80 milliliters per minute per 1.73 meter^2 (ml/min/1.73 m^2) during screening (using the Chronic Kidney Disease Epidemiology Collaboration formula)
  4. History or current evidence of ongoing hepatic disease or impaired hepatic function at screening.
  5. A participant will be excluded if more than one of the following lab value deviations are found: 1) aspartate transaminase (AST) (>= 1.2 upper limit of normal [ULN]), alanine transaminase (ALT) (>=1.2 ULN), 2) gamma-glutamyl transpeptidase (GGT) (>=1.2 ULN), alkaline phosphatase (ALP) (>=1.2 ULN), 3) total bilirubin (>2.00 milligrams per deciliter [mg/dL]) or creatine kinase (>=3 ULN). A single deviation from the above values is acceptable and will not exclude the participant, unless specifically advised by the investigator, or medically qualified designee;
  6. Evidence of urinary obstruction (example, due to benign prostate hyperplasia) or difficulty in voiding at screening;
  7. History or clinical evidence (on physical examination) at screening of pancreatic injury or pancreatitis.
* Any vaccination, including Coronavirus disease (COVID)-19 vaccine, within 14 days prior to the first dose.
* History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to dosing.
* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 milliliters (mL) of beer 5 percent (%), 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* Positive urine drug screen or urine alcohol test at screening or Day -1.
* Positive cotinine test at screening or Day -1
* Participant reported regular consumption of beverages or food containing xanthine derivatives or xanthine-related compounds (example, coffee, tea, caffeine-containing sodas and chocolate), equivalent to >= 500 milligrams (mg) xanthine per day.
* Current smoker, defined as the use of tobacco or nicotine products during the 3 months prior to screening until admission to the unit.
* Participant reports consumption of any drug metabolizing enzyme (example, Cytochrome P450 3A4 [CYP3A4] or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (example, broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort etcetera [etc.]) within 2 weeks prior to admission to the unit.
* Positive results in any of the serology tests for human immunodeficiency virus (HIV) antigen (Ag) and antibody (Ab), Hepatitis C virus antibody (HCV-Ab), hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) (immunoglobulin [Ig]G + IgM).
* Performance of strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission and does not agree to refrain throughout the entire study.
* Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the Investigator's or medically qualified designee's opinion may pose a risk to the participant.
* Any condition not identified in the protocol that in the opinion of the investigator or medically qualified designee would confound the evaluation and interpretation of the study data or may put the participant at risk.
* Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
* Hemoglobin value <12.0 grams per deciliter [g/dL] for males and <11.5 g/dL for females, may repeat at discretion of the Investigator or medically qualified designee at screening or day -1.
* Participant who has previously been enrolled in this study.
* Participant has unsuitable veins for multiple venipunctures/cannulations as assessed by the investigator or delegate at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Post-dose Concentration (Cmax) for Ibuprofen Under Fasted Conditions (ADA Liquid Filled Capsules [Treatment A] vs. ADA Caplet [Treatment B]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cmax is defined as the maximum observed post-dose concentration for ibuprofen obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
Area Under the Plasma Concentration Versus Time Curve Calculated from Time 0 to the Last Measurable Sampling Time Point, t (AUC[0-t]) for Ibuprofen Under Fasted Conditions (ADA Liquid Filled Capsules [Treatment A] vs. ADA Caplet [Treatment B]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
Cmax for Acetaminophen Under Fasted Conditions (ADA Liquid Filled Capsules [Treatment A] vs. ADA Caplet [Treatment B]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cmax is defined as the maximum observed post-dose concentration for acetaminophen obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
AUC(0-t) for Acetaminophen Under Fasted Conditions (ADA Liquid Filled Capsules [Treatment A] vs. ADA Caplet [Treatment B]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
Cmax for Ibuprofen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cmax is defined as the maximum observed post-dose concentration for ibuprofen obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
AUC(0-t) for Ibuprofen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to Infinity (AUC[0-inf]) for Ibuprofen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).
Cmax for Acetaminophen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cmax is defined as the maximum observed post-dose concentration for acetaminophen obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
AUC(0-t) for Acetaminophen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
AUC(0-inf) for Acetaminophen (ADA Liquid Filled Capsules Under Fed Conditions [Treatment C] vs. ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A]) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).

SECONDARY OUTCOMES:
Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  %AUCex is defined as the percentage of AUC(0-inf) obtained by extrapolation, calculated as (1-[AUC0-t/AUC0-inf]) *100. Blood samples will be collected at indicated timepoints for the analysis of %AUCex.
AUC(0-inf) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).
Terminal Elimination Rate Constant (λz) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  λz is defined as the terminal elimination rate constant computed as the negative of the slope of the regression line of ln(C[t]) on time. Blood samples will be collected at indicated timepoints for the analysis of λz.
Time of the Maximum Observed Post-dose Concentration (tmax) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Blood samples will be collected at indicated timepoints for the analysis of tmax.
Elimination Half-life (t1/2) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  t1/2 is defined as the elimination half-life computed as t1/2 = ln(2)/λz where λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of t1/2.
Apparent Volume of Distribution (Vz/F) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Vz/F is defined as the apparent volume of distribution, as calculated by the dose administered/(λz *AUC0-inf) where λz is the terminal elimination rate constant and AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Vz/F.
Apparent Total Clearance (Cl/F) for Ibuprofen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cl/F is defined as the apparent total clearance, as calculated by the dose administered/AUC0-inf where AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Cl/F.
%AUCex for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  %AUCex is defined as the percentage of AUC(0-inf) obtained by extrapolation, calculated as (1-[AUC0-t/AUC0-inf]) *100. Blood samples will be collected at indicated timepoints for the analysis of %AUCex.
AUC(0-inf) for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).
λz for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  λz is defined as the terminal elimination rate constant computed as the negative of the slope of the regression line of ln(C[t]) on time. Blood samples will be collected at indicated timepoints for the analysis of λz.
tmax for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Blood samples will be collected at indicated timepoints for the analysis of tmax.
t1/2 for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  t1/2 is defined as the elimination half-life computed as t1/2 = ln(2)/λz where λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of t1/2.
Vz/F for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Vz/F is defined as the apparent volume of distribution, as calculated by the dose administered/(λz *AUC0-inf) where λz is the terminal elimination rate constant and AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Vz/F.
Cl/F for Acetaminophen (Treatment A, Treatment C, Treatment B and Treatment D) | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cl/F is defined as the apparent total clearance, as calculated by the dose administered/AUC0-inf where AUC(0-inf) is the area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples will be collected at indicated timepoints for the analysis of Cl/F.
Cmax for Ibuprofen (ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A] vs. Advil Liqui-gel Under Fasted Conditions [Treatment D] | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  Cmax is defined as the maximum observed post-dose concentration for ibuprofen obtained without interpolation. Blood samples will be collected at indicated timepoints for the analysis of Cmax.
AUC(0-t) for Ibuprofen (ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A] vs. Advil Liqui-gel Under Fasted Conditions [Treatment D] | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-t) is defined as the area under the plasma concentration versus time curve calculated from time 0 to the last measurable sampling time point, t, computed using the linear trapezoidal rule. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-t).
AUC(0-inf) for Ibuprofen (ADA Liquid Filled Capsules Under Fasted Conditions [Treatment A] vs. Advil Liqui-gel Under Fasted Conditions [Treatment D] | Pre-dose (within 1 hour prior to dosing) and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.5, 6, 8,10,12,16,20, and 24 hours post dose on Day 1 in each treatment period (each period is of 3 days)
  AUC(0-inf) is defined as the area under the plasma concentration versus time curve calculated from time 0 to infinity. AUC(0-inf) = AUC(0-t) + C(t)/λz where C(t) is the concentration at the last measurable sampling time point and λz is the terminal elimination rate constant. Blood samples will be collected at indicated timepoints for the analysis of AUC(0-inf).
Number of Participants Reporting Ease of Swallowing: Categorical Response | Post Dose on Day 1 in each treatment period (each period is of 3 days)
  Immediately after dosing, participants will be asked to evaluate the ease of swallowing to assess the acceptability of each treatment. Participants will be asked to provide a categorical response (Agree/Disagree) to the question "Do you agree or disagree that the product is Easy to swallow?". Number of participants providing response to the question will be reported.
Number of Participants Reporting Ease of Swallowing on a 5-Point Ordinal Scale | Post Dose on Day 1 in each treatment period (each period is of 3 days)
  Immediately after dosing, participants will be asked to rank the ease of swallowing of each product on a 5-point ordinal scale with scores ranging from 1 to 5 where 1=not easy to swallow; 2=somewhat easy to swallow; 3=average to swallow; 4=above average to swallow; 5=very easy to swallow. Higher score indicates more ease in swallowing.

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.